CLINICAL TRIAL: NCT03366155
Title: A Single-Arm Phase II Study of Hepatic Artery Infusion Pump Chemotherapy With Floxuridine and Dexamethasone in Combination With Systemic Chemotherapy for Patients With Colorectal Cancer Metastatic to the Liver
Brief Title: Hepatic Artery Infusion Pump Chemotherapy With Floxuridine and Dexamethasone in Combination With Systemic Chemotherapy for Patients With Colorectal Cancer Metastatic to the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180024; 18-C-0024
Record Dates: First submitted 2017-12-07; First posted 2017-12-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01-06

CONDITIONS: Colorectal Cancer; Liver Metastases; Colorectal Adenocarcinoma; Colorectal Cancer With Hepatic Metastases; Colorectal Carcinoma
Keywords: Unresectable Liver Tumor; Response Rates; Progression-Free Survival; Patient Survival
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Oxaliplatin; Fluorouracil; Irinotecan; Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/ Arm 1 (Experimental): HAIP chemotherapy + Systemic chemotherapy
  Interventions: Device: Codman 3000 constant flow pump catheter; Drug: Panitumumab; Drug: FUDR-Dex; Drug: Oxaliplatin; Drug: 5FU; Drug: Irinotecan; Procedure: HAIP installation; Drug: cetuximab; Device: Medtronic SynchroMed II Pump

INTERVENTIONS:
Device: Codman 3000 constant flow pump catheter — implanted Medtronic SynchroMed II Pump with codman 3000 Constant Flow Pump Catheter
Drug: Panitumumab — 6 mg/kg, IV
Drug: FUDR-Dex — HAIP will be filled with mixture of Floxuridine and Dexamethasone. Pump will perfuse drugs to liver for 14 days. Floxuridine (0.12 mg/kg X pump volume X pump flow rate),Dexamethasone (1 mg/day X pump volume (30) X pump flow rate)
Drug: Oxaliplatin — 85 mg/m2, IV
Drug: 5FU — 2000 mg/m2, IV 46-hour infusion of 5-Fluorouracil + 400 mg/m2, IV of Leucovorin
Drug: Irinotecan — 150 mg/m2, IV
Procedure: HAIP installation — HAI pump installation
Drug: cetuximab — 500 mg/m2, IV
Device: Medtronic SynchroMed II Pump — implanted Medtronic SynchroMed II Pump with Codman 3000 Constant Flow Pump Catheter

SUMMARY:
Background:

Many people with colorectal cancer get liver metastases. Standard treatment for this is a combination of chemotherapy drugs. Directing the chemotherapy to the liver may be effective. A device that does this a pump that delivers drugs over 2 weeks at constant rate into the hepatic artery. The person s body temperature causes the drug to flow from the pump. Researchers want to see if this helps people with colorectal metastases to the liver.

Objective:

To study the effectiveness of a hepatic artery infusion pump at treating colorectal metastases to the liver.

Eligibility:

Adults at least 18 years old with colorectal metastases to the liver

Design:

Participants will be screened with:

Medical history

Physical exam

Heart, blood, and urine tests

Scans

Participants will stay in the hospital a few days. A small plastic tube (catheter) will be inserted in an artery into the liver. The catheter will be attached to the pump. That will lie under the skin on the abdomen. It will be small and participants will be able to feel it.

Participants will get treatment in 28-day cycles.

Every Day 1, they will have physical exam, symptom review, and blood tests.

Every 2 weeks, they will come to the clinic to get chemotherapy by a catheter or port.

Every 12 weeks, they will have a scan.

Tissue samples may be taken during the study.

When they finish the drug, participants may have the pump removed. They will repeat the Day 1 tests. They will be called every 6 months to see how they are doing.

DETAILED DESCRIPTION:
Background:

* Nearly 60% of patients with colorectal cancers will develop liver metastases over the course of their disease.
* Of patients with metastatic colorectal cancer, the liver will be the sole site of recurrence or the survival-limiting site of disease for 20%.
* Liver directed therapy, which has taken many forms over the last several decades, is a potential means to prolong survival for properly selected patients and delay progression at that site.
* Hepatic artery infusion of floxuridine (FUDR) via an implantable hepatic artery infusion pump (HAIP) induces objective clinical response rates of nearly 50% in heavily pre-treated patients with metastatic colorectal cancer to the liver.
* The identification of patients likely to respond to HAIP and those likely to suffer pumprelated adverse events is currently unknown, and has limited the wide-spread adoption of this otherwise well tolerated intervention.

Objective:

* To assess the safety of hepatic artery infusion therapy using the Medtronic pump with the Codman catheter.
* To determine the response rate in patients with unresectable metastatic colorectal cancer treated with HAIP chemotherapy as measured by RECIST.

Eligibility:

* Histologically or cytologically confirmed colorectal adenocarcinoma metastatic to the liver.
* Patients with liver metastases not amenable to resection to No Evidence of Disease (NED) in one stage.
* Patients must have received systemic chemotherapy.
* Age greater than or equal to 18 years.

Design:

- Single arm, Phase II study of HAIP chemotherapy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed diagnosis of colorectal adenocarcinoma.
* Patients must have measurable liver metastatic disease.
* Patients must have progressed on, been intolerant of or have residual disease after oxaliplatin- or irinotecan-containing, fluorouracil-based, chemotherapeutic regimen.
* Age greater than or equal to 18 years.
* ECOG performance status less than or equal to 1
* Patients must have adequate organ and marrow function as defined below:

  * leukocytes > 3,000/mcL
  * absolute neutrophil count > 1,500/mcL
  * platelets > 90,000/mcL
  * total bilirubin < 1.5 X institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR eGFR within normal as predicted by the CKD-EPI equation > 60 mL/min/1.73 m2.
* The hepatic artery infusion pump chemotherapy has potential teratogenic and/or abortifacient effects. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and after completion of study treatment : 3 months after the last study drug for men; 6 months after the last study drug for women. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Arterial anatomy on CT angiogram amenable to placement of the HAIP.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* HIV-positive patients may be considered for this study only after consultation with an HIV trained physician.
* Patients must agree to co-enroll on the Surgical Oncology Program s tissue collection protocol 13C0176, 'Tumor, Normal Tissue and Specimens from Patients Undergoing Evaluation or Surgical Resection of Solid Tumors'

EXCLUSION CRITERIA:

* Patients with liver metastases amenable to resection to No Evidence of Disease (NED) in one stage.
* Patients who are receiving any other investigational agents.
* Patients with incontrovertible radiographic evidence of disease outside of the colon/rectum (primary) and liver given unlikelihood of benefit from liver-directed therapy.

Note: The exception to this exclusion is patients with fewer than five lung lesions greater than 1 cm that have not increased in size by more than 10% over a 4-month period of time, and are amenable to resection should subsequent problematic growth occur. Lesions less than 1 cm are indeterminant as far as etiology is concerned and will be ignored. Patients with liver metastases and oligometastatic lung lesions (we define oligometastatic as less than 5 amenable to thoracoscopic removal) are still likely to benefit from liver directed therapy.

* Patients who have undergone extra-hepatic metastasectomy and have a documented disease-free interval less than or equal to 4 months.
* MSI-high patients who need to be treated with check-point inhibitors
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. This also includes any condition, including the presence of laboratory abnormalities, which in the opinion of the Principal Investigator places the subject at unacceptable risk if they were to participate in the study or confounds the ability to interpret data from the study.
* Active concurrent malignancies within the last five years other than colorectal primary except basal cell skin carcinoma and thyroid carcinoma.
* Prior radiation to liver.
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects of the HAIP chemotherapy. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with HAIP, breast-feeding should be discontinued if the mother is treated. These potential risks may also apply to other agents used in this study. Lactating women must-not breastfeed during study treatment and until at least 7 days after the final dose of study drug(s).
* Patients with active Hepatitis B or C infection because of the potential for increased liver toxicity given the damaging effects of the virus.
* History of allergic reactions attributed to compounds of similar chemical composition to FUDR or heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) | at progression
  The fraction of patients who experience a PR or CR using the study treatment

SECONDARY OUTCOMES:
Overall survival | death
  Median amount of time subject survives after therapy
Hepatic progression-free survival | at progression
  The fraction of patients whose tumors in liver shrunk after therapy
Extra-hepatic progression-free survival | at progression
  The fraction of patients whose tumors outside liver shrunk after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Hernandez, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Ammori JB, Kemeny NE, Fong Y, Cercek A, Dematteo RP, Allen PJ, Kingham TP, Gonen M, Paty PB, Jarnagin WR, D'Angelica MI. Conversion to complete resection and/or ablation using hepatic artery infusional chemotherapy in patients with unresectable liver metastases from colorectal cancer: a decade of experience at a single institution. Ann Surg Oncol. 2013 Sep;20(9):2901-7. doi: 10.1245/s10434-013-3009-3. Epub 2013 Jun 15. PMID 23771246
- [Background] D'Angelica MI, Correa-Gallego C, Paty PB, Cercek A, Gewirtz AN, Chou JF, Capanu M, Kingham TP, Fong Y, DeMatteo RP, Allen PJ, Jarnagin WR, Kemeny N. Phase II trial of hepatic artery infusional and systemic chemotherapy for patients with unresectable hepatic metastases from colorectal cancer: conversion to resection and long-term outcomes. Ann Surg. 2015 Feb;261(2):353-60. doi: 10.1097/SLA.0000000000000614. PMID 24646562
- [Background] Cercek A, D'Angelica M, Power D, Capanu M, Gewirtz A, Patel D, Allen P, Fong Y, DeMatteo RP, Jarnagin WR, Kemeny NE. Floxuridine hepatic arterial infusion associated biliary toxicity is increased by concurrent administration of systemic bevacizumab. Ann Surg Oncol. 2014 Feb;21(2):479-86. doi: 10.1245/s10434-013-3275-0. Epub 2013 Oct 24. PMID 24154839
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0024.html